CLINICAL TRIAL: NCT04191161
Title: Efficacy of Lumbar Immobilisation by Rigid Brace for Chronic Low Back Pain Patients With Modic 1 Changes
Brief Title: Efficacy of Lumbar Immobilisation by Rigid Brace for Chronic Low Back Pain Patients With Modic 1 Changes (DICO)
Acronym: DICO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2019 COUDEYRE; 2019-A00861-56 (Other: ANSM)
Record Dates: First submitted 2019-12-06; First posted 2019-12-09 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Chronic Pain
Keywords: Modic type I; Chronic low back pain; Rigid brace
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Patients will be recruited if aged between 18 and 55 years old and suffering from chronic lumbar pain (Visual Analogic Scale (VAS) > 3) associated with Modic type I changes diagnosed with a MRI achieved less than 6 months before the consultation and interpreted by a radiologist specialised in spine disease. Patients must also be capable of giving a clear consent. Will not be included patients suffering from other types of Modic change, or any other cause of back pain such as spondylolisthesis, fracture, spondylitis, scoliosis, rheumatoid arthritis and also patient not willing to wear the brace for at least 3 months. Patients will be recruited from the consultation in PMR units across 5 centres in France.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brace group (Experimental): patients will receive their brace 2 weeks after the first consultation (usual delay to conceive and deliver the brace), they will be asked to wear the brace all day and will be allowed to redraw it at night. Brace must be worn for 3 months. A specific eduction on how to wear the brace will also be delivered. A thermal sensor chip will be placed in the brace to assess the observance. No physiotherapy will be prescribed during this period. Patient will attend to 3 consultations, day 0, 3 months and finally at 6 months later. These three consultations are part of usual care.
  Interventions: Device: Wearing the rigid brace
- Control group (Placebo Comparator): patients will continue physiotherapy sessions if already prescribed but no extra sessions will be prescribed. Pain killers will be adjusted. Patients will also attend to three consultations such as described above. Main outcome will be assessed at M3. After M3, patients who did not receive the brace will have the choice to receive it for the next 3 months and secondary outcome will be assessed at 6 months.
  Interventions: Device: Wearing the rigid brace

INTERVENTIONS:
Device: Wearing the rigid brace — Custom braces are made from 4mm thick polyethylene with Velcro® fastening. They are Computer Aided Designed and are made by the same manufacturer (LAGARRIGUE). A thermal sensor chip will placed in the brace to assess observance.

SUMMARY:
Chronic low back pain may be associated with active discopathy. This subset of individuals are defined by a clinical and radiological syndrome with specific MRI signals, known as MODIC changes.

Three types (I, II and III) of MODIC changes are described. Type I refers to the inflammatory reaction regarding the intervertebral-disc subchondral bone and adjacent vertebral-endplate subchondral bone. The natural evolution of this active discopathy will lead to sclerosis (type III) supposedly less painful. So far the underlying mechanism remains unclear and debated (mechanical, local infection, genetic). In the absence of international guidelines on the management on chronic low back pain with MC type 1, different therapeutic strategies have been described. The main goal is to accelerate the transition to MC type 2, which is supposedly less painful. The estimated time to expect a transition from type 1 to type 2 is at least 1 year.

The mechanical hypothesis found its origin in the Modic et al. initial study, linking Modic changes (MC) types 1 and 2 to degenerative disc disease.

The Histological analysis of patient suffering from active discopathy has shown signs of micro fractures regarding vertebral endplates. The local inflammatory reaction may be part of a repair process following the micro fracture. Based on this mechanical explanation an orthopaedic treatment with a lumbar brace may accelerate the healing, thus the transition from modic I to type II. This approach has been studied in a retrospective analysis on 62 patients suffering from active discopathy (modic type I) who were prescribed a custom lumbar rigid brace for 3 months, at endpoint 80% of the patients treated described a reduction of at least 30% of their initial pain.

This study aims to confirm the previous hypothesis, that lumbar immobilisation by custom rigid brace can reduce the pain after being worn for 3 months. Secondary objective will be to assess the pain reduction at 6 months along with functional outcome, fears and beliefs, mood and medical costs at short (3 months) and mid (6months) term.

DETAILED DESCRIPTION:
This will be a 2 parallel group multicentre randomised controlled trial. Patients will undergo 3 consultations with the physician, based on the usual follow up for this pathology. During the first consultation the physician will check the inclusion criteria, medical history, clinical data relative to the different outcomes, and prescribe optimizated pain killers and deliver information about self care and physical activity. Patient reported outcome measures will be assessed through self answering questionnaires with the help of a research assistant if necessary. After randomisation the prosthetist will take the measurement to conceive the custom brace. Patients will then be re-examined during a 2nd consultation 3 month later to assess the main outcome (pain reduction) and other secondary outcome (proms). A third consultation will be organised 6 months later for secondary outcome (pain reduction and proms).

ELIGIBILITY:
Inclusion Criteria:

-- Age: > 18 years < 55 years

* Patient affiliated to a social security scheme ( beneficiary entitled )
* Patient has given its consent in writing to participate in the study
* Low back pain associated with a MODIC I signal at the lumbar stage objectified by an MRI dated less than 6 months and confirmed by a radiologist.

Exclusion Criteria:

* Other types of Modic change
* Other cause of back pain such as spondylolisthesis, fracture, spondylitis, scoliosis, rheumatoid arthritis and also
* Patient not willing to wear the brace for at least 3 months
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Reduction of the pain intensity | Month 3
  Average change from baseline in the pain intensity measured on a Visual Analogical Scale (VAS) Visual analog scale (VAS) and its corresponding visual analog pain scale, is a psychometric scale that is generally used to conduct pain scale surveys to understand varying degrees of pain or discomfort experienced by a patient. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm)

SECONDARY OUTCOMES:
The Roland Morris Disability Questionnaire measures in patients with low back pain | Month 3
  The Roland-Morris Questionnaire is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale. The RMQ has been shown to yield reliable measurements, which are valid for inferring the level of disability, and to be sensitive to change over time for groups of patients with low back pain. Roland and Morris did not provide descriptions of the varying degrees of disability (eg, 40%-60% is severe disability). Clinical improvement over time can be graded based on the analysis of serial questionnaire scores. If, for example, at the beginning of treatment, a patient's score was 12 and, at the conclusion of treatment, their score was 2 (10 points of improvement), we would calculate an 83% (10/12 x 100) improvement
The Roland Morris Disability Questionnaire measures in patients with low back pain | Month 6
  The Roland-Morris Questionnaire is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale. The RMQ has been shown to yield reliable measurements, which are valid for inferring the level of disability, and to be sensitive to change over time for groups of patients with low back pain. Roland and Morris did not provide descriptions of the varying degrees of disability (eg, 40%-60% is severe disability). Clinical improvement over time can be graded based on the analysis of serial questionnaire scores. If, for example, at the beginning of treatment, a patient's score was 12 and, at the conclusion of treatment, their score was 2 (10 points of improvement), we would calculate an 83% (10/12 x 100) improvement
The fears and beliefs measured by questionnaire FABQ | Month 3
  The FABQ can help predict those that have a high pain avoidance behavior. Clinically, these people may need to be supervised more than those that confront their pain. The FABQ contains 2 scales: a work scale (FABQ-W) composed of 7 items and a physical activity scale (FABQ-PA) composed of 4 items. The two scales are scored separately. Higher FABQ scores indicate elevated fear-avoidance beliefs. "FABQ-W" has a point score that ranges from 0-42 points. It can be calculated as follows: (Total points for items 6, 7, 9, 10 11, 12 and 15) = Work scale score. "FABQ-PA" can range from 0-24 points. Scores are calculated as follows: (Total points for items 2, 3, 4 and 5) = Physical activity scale score.
The fears and beliefs measured by questionnaire FABQ | Month 6
  The FABQ can help predict those that have a high pain avoidance behavior. Clinically, these people may need to be supervised more than those that confront their pain. The FABQ contains 2 scales: a work scale (FABQ-W) composed of 7 items and a physical activity scale (FABQ-PA) composed of 4 items. The two scales are scored separately. Higher FABQ scores indicate elevated fear-avoidance beliefs. "FABQ-W" has a point score that ranges from 0-42 points. It can be calculated as follows: (Total points for items 6, 7, 9, 10 11, 12 and 15) = Work scale score. "FABQ-PA" can range from 0-24 points. Scores are calculated as follows: (Total points for items 2, 3, 4 and 5) = Physical activity scale score.
The knowledge of emotional state measured by questionnaire HAD (Hospital Anxiety and Depression) | Month 3
  The Hospital Anxiety and Depression Scale (HADS) is a valid and reliable self-rating scale that measures anxiety and depression in both hospital and community settings. HADS gives clinically meaningful results as a psychological screening tool and can assess the symptom severity and caseness of anxiety disorders and depression in patients with illness and the general population.
  * One questionnaire, comprising fourteen questions. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
  * Scoring : 0-7- normal, 8-10-borderling abnormal, 11-21-abnormal
The knowledge of emotional state measured by questionnaire HAD (Hospital Anxiety and Depression) | Month 6
  The Hospital Anxiety and Depression Scale (HADS) is a valid and reliable self-rating scale that measures anxiety and depression in both hospital and community settings. HADS gives clinically meaningful results as a psychological screening tool and can assess the symptom severity and caseness of anxiety disorders and depression in patients with illness and the general population.
  * One questionnaire, comprising fourteen questions. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
  * Scoring : 0-7- normal, 8-10-borderling abnormal, 11-21-abnormal
Patient Global Impression of Change by Scale PGIC | Month 3
  This scale evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status. It consists of one item. Patient choose: 1 -No change (or condition has gotten worse), 2 - Almost the same, hardly any change at all, 3 - A little better, but no noticeable change, 4 - Somewhat better, but the change has not made any real difference, 5 - Moderately better, and a slight but noticeable change, 6 - Better and a definite improvement that has made a real and worthwhile difference, 7 - A great deal better and a considerable improvement that has made all the difference.
Patient Global Impression of Change by Scale PGIC | Month 6
  This scale evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status. It consists of one item. Patient choose: 1 -No change (or condition has gotten worse), 2 - Almost the same, hardly any change at all, 3 - A little better, but no noticeable change, 4 - Somewhat better, but the change has not made any real difference, 5 - Moderately better, and a slight but noticeable change, 6 - Better and a definite improvement that has made a real and worthwhile difference, 7 - A great deal better and a considerable improvement that has made all the difference.
patient preference towards the treatment received | day 0
  question asked by investigator to patient
medical costs | month 3
  social security expenses such brace price, number of physiotherapy sessions, sick leave duration, pharmacologic treatment, consultations linked to chronic low back pain (general practitioner or specialist) and complementary examination (MRI, CT scans, radiography, blood analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Coudeyre, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France